CLINICAL TRIAL: NCT05040022
Title: Quality of Recovery After Laparoscopic Cholecystectomy Under Moderate Neuromuscular Blockade Using Low Pressure or Standard Pneumoperitoneum Pressure
Brief Title: Quality of Recovery Under Low or Standard Pneumoperitoneum Pressure
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Pontificia Universidade Catolica de Sao Paulo (Other)
Responsible Party: Principal Investigator, Eduardo Toshiyuki Moro, Professor, Pontificia Universidade Catolica de Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CAAE 49753621.1.0000.5373
Record Dates: First submitted 2021-09-02; First posted 2021-09-10 (Actual); Last update posted 2021-09-20 (Actual); Status verified 2021-09

CONDITIONS: Quality of Recovery; Postoperative Pain; Postoperative Nausea and Vomiting; Neuromuscular Blockade
MeSH Terms: conditions — Pain, Postoperative; Postoperative Nausea and Vomiting

STUDY DESIGN:
Intervention Model Description: Prospective, randomized and double-blinded
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Patients will be randomized according to the sequence of random numbers generated by a computer using a specific program (www.random.org). For each patient, an opaque envelope containing the group to which the patient will be allocated will be prepared, sealed, and numbered sequentially.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group pneumoperitoneum pressure 10 (Active Comparator): Pneumoperitoneum pressure at 10 mmHg
  Interventions: Drug: Pneumoperitoneum pressure 10 mmHg
- Group neumoperitoneum pressure 14 (Placebo Comparator): Pneumoperitoneum pressure at 10 mmHg
  Interventions: Drug: Pneumoperitoneum pressure 14 mmHg

INTERVENTIONS:
Drug: Pneumoperitoneum pressure 10 mmHg — The abdomen will be inflated with carbon dioxide to maintain the intra-abdominal pressure at 10 mmHg (group 10)
  Arms: Group pneumoperitoneum pressure 10
Drug: Pneumoperitoneum pressure 14 mmHg — The abdomen will be inflated with carbon dioxide to maintain the intra-abdominal pressure at 14 mmHg (group 14).
  Arms: Group neumoperitoneum pressure 14

SUMMARY:
The use of low-pressure pneumoperitoneum seems to be able to reduce complications such as postoperative pain. However, the quality of evidence for most studies evaluating this relationship is considered low. The absence of concealment of pneumoperitoneum pressure and the lack of description of neuromuscular blockade characteristics are the main causes of bias. The purpose of this study will be to evaluate by means of a prospective, randomized and double-blinded trial, the quality of recovery (QoR-15) questionnaire of patients undergoing laparoscopic cholecystectomy under moderate neuromuscular blockade, using low pneumoperitoneum pressure or "standard" pressure. Eighty patients submitted to laparoscopic cholecystectomy and randomly distributed in two groups will be included: low pneumoperitoneum pressure (10 mmHg) or "standard" pressure (14 mmHg). The value of abdominal pressure will be kept hidden for all participants, except for the nurse responsible for the operating room. Moderate neuromuscular blockade will be maintained according to Train-of-four count (TOFc) = 3 for all cases.

DETAILED DESCRIPTION:
METHODS After obtaining approval from the Research Ethics Committee of the Faculty of Medical and Health Sciences of PUC-SP on August 10th 2021, CAAE 49753621.1.0000.5373, patients 18 to 70 years of age, with physical status I and II according to the American Society of Anesthesiologists (ASA), undergoing elective laparoscopic cholecystectomy at Hospital Santa Lucinda will be evaluated for participation in this clinical, prospective, and randomized clinical trial. Patients will be excluded before randomization if: (i) refuse to participate; (ii) present inability to communicate due to altered level of consciousness or due to the presence of neurological or psychiatric illness; (iii) present contraindication to the use of any of the drugs employed in the study; (iv) present history of alcohol or drug addiction; (v) body mass index (BMI) ≥ 35; (vi) and the presence of chronic pain or use of opioids.

Study sequence

Patients will be randomized according to the sequence of random numbers generated by a computer using a specific program (www.random.org). For each patient, an opaque envelope containing the group to which the patient will be allocated will be prepared, sealed, and numbered sequentially. On the day of the surgery, after the pre-anesthetic evaluation and the necessary explanation about the study, study consent will be obtained. Age, gender, physical status, body mass index (BMI) and risk classification for post-operative nausea and vomiting (PONV) will be recorded as proposed by Apfel et al. All patients will be instructed on the numerical scale of post-operative pain and on the QoR-15 questionnaire. No pre-anesthetic medication will be administered.

Anaesthesia and surgery After entering the operating room, all patients will be monitored with ASA standard monitoring. NMB will be assessed using acceleromyography (TOF Watch SX®; Schering-Plow) as recommended for use in clinical research. The acceleration transducer will be attached to the volar side in the distal phalanx of the thumb. Anaesthesia will be induced using 0.5 µg/kg remifentanil for 3 minutes, followed by propofol (2 mg/kg), and rocuronium (0.3 mg/Kg). After tracheal intubation anesthesia will be maintained with 1.5%-3% sevoflurane and 0.1-0.5 µg/kg/min remifentanil, both necessary to maintain an adequate anesthesia plane. The ventilation will be controlled with the tidal volume and respiratory rate adjusted aiming for an end-tidal CO2 between 30 and 40 mmHg. Additional doses of rocuronium (0.05 mg/kg) will be administered to maintain TOFc = 3 until gallbladder removal. TOF stimulation will be applied every 15 minutes and the time under moderate or deep NMB will be registered. Hydration will be achieved using lactated Ringer's solution (500 ml in the first 30 minutes followed by 2 ml/kg/h maintenance). All patients will receive dexamethasone (8 mg) and ketoprofen (100 mg) at the beginning of the surgery and ondansetron (4 mg) 15 minutes before the end of the procedure. Atropine (0.02 mg/kg) and neostigmine (0.05 mg/kg) will be administered to obtain T4/T1 > 0.9 and, after awakening, extubation will be performed. The time elapsed between the discontinuation of the anesthetic agents and awakening will be recorded. Furthermore, the duration of the surgery and the total dose of rocuronium will be noted. Local anesthetic infiltration of the trocar insertion sites will be performed by the surgical team using 20 ml of 0.75% ropivacaine under direct visualization, and included the aponeurosis, the subcutaneous tissue, and the skin. The abdomen will be inflated with carbon dioxide to maintain the intra-abdominal pressure at 10 mmHg (group 10) or 14 mmHg (group 14). The display of the insufflation pressure value was blinded to the surgical team and the anesthesiologist, but not the operating room nurse. At the end of surgery, irrigation of the abdominal cavity and the surgical site will be performed using saline solution. The pneumoperitoneum will be completely decompressed in all patients using manual compression. Surgery will be performed by the same surgical team comprised of two experienced laparoscopists and two resident clinicians. At the end of the procedure, the surgical team will be asked to classify the surgical conditions (good visualization, adequate working space) using a 5-point Likert scale of 'very bad' (1) to 'excellent' (5). The patients will be transferred to the PACU and monitored until the criterion for discharge were met (score according to the Aldrete and Kroulik modified scale = 10). During the PACU stay, the magnitude of pain, nausea, vomiting, and PACU length of stay will be documented. Pain will be evaluated every 15 minutes using a verbal numeric scale (VNS) of 0-10, where 0 was 'no pain' and 10 the 'most severe pain imaginable'. Intravenous morphine will be administered every 5 minutes to obtain a score <3 (2 mg for pain <7 and 3 mg for pain ≥7). PONV will be treated with intravenous dimenhydrinate 30 mg. Following PACU discharge to the ward, patients will receive 100 mg of ketoprofen every 12 hours and 1 g of dipyrone every 6 hours intravenously. Whenever the patient considers the analgesic regimen to be insufficient, tramadol 100 mg will be administered orally at intervals of up to 8 hours. In case of nausea and/or vomiting, ondansetron 8 mg will be administered intravenously. Pain intensity (VNS) will be recorded at 4, 8, 12 and 24 hours after arrival on the ward. Tramadol utilization as well as the occurrence of nausea, vomiting and other complications will be documented. As per institutional protocol, all study patients remain in hospital for a period of 24 hours.

Questionnaire QoR-15 The interviews will be conducted: immediately after opening the envelope that will define the group in which the patient will be included. The preoperative questionnaire (QoR-15) will be applied by a physician of the residency program in anesthesiology and, after surgery, by one of three medical students, unrelated to the anesthetic procedure performed. The QoR-15 has 15 questions divided into 5 dimensions: emotional state, physical comfort, psychological support, physical independence and pain. Each question should generate a score based on a numerical scale of 11 points (zero to 10), totaling zero (poor recovery) up to 10 (excellent recovery).

Statistical analysis The sample size was calculated considering a power of 90% to detect a difference of 8 points in the QoR-15, which indicates the need to include 35 participants in each group. Considering possible losses, the final sample will include 80 patients.

ELIGIBILITY:
Inclusion Criteria:

* Physical status I and II according to the American Society of Anesthesiologists (ASA)
* Undergoing elective laparoscopic cholecystectomy

Exclusion Criteria:

* refuse to participate
* Present inability to communicate due to altered level of consciousness or due to the presence of neurological or psychiatric illness
* Present contraindication to the use of any of the drugs employed in the study
* Present history of alcohol or drug addiction
* Body mass index (BMI) ≥ 35
* Presence of chronic pain or use of opioids.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-10-01 (Estimated); Primary Completion 2022-01-05 (Estimated); Study Completion 2022-01-15 (Estimated)

PRIMARY OUTCOMES:
Quality of recovery | From randomization up to 15 days
  The quality of recovery will be assessed using the Qualtity of Recovery 15
  questionnaire. Total scores range from 0 to 150. Higher scores mean a better outcome.

SECONDARY OUTCOMES:
Postoperative pain | From the PACU arriving up to 24 hours
  Pain intensity (Verbal Numeric Scale) will be assessed at 15, 30, 45 and 60 minutes during postanesthetic unit (PACU) stay and 4, 8, 12 and 24 hours after arrival on the ward.Verbal Numeric Scale scores range from 0 to 10. Higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Moro, Principal Investigator — Faculdade de Ciências Médicas e da Saúde PUCSP
Locations (1):
- Eduardo T Moro, Araçoiaba da Serra, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Results will be submitted to publication
Supporting Information: Study Protocol, SAP
Time Frame: When summary data are published
Access Criteria: The access will be related to the journal (open access or not)